CLINICAL TRIAL: NCT01195493
Title: Clinical and Microbiological Effects of an Essential Oils Solution Used as an Adjunct to Daily Oral Hygiene Practices in Chronic Periodontitis Patients in Supportive Care
Acronym: Listerine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2009/552
Record Dates: First submitted 2010-09-03; First posted 2010-09-06 (Estimated); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Chronic Periodontitis
Keywords: Chronic periodontitis
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- test mouthrinse (Experimental)
  Interventions: Other: Essential Oils solution
- control group (Active Comparator)
  Interventions: Other: negative control solution

INTERVENTIONS:
Other: Essential Oils solution — (Essential oils solution, Listerine®, Johnson & Johnson) to use twice a day (2 x 20 ml) following daily mechanical oral hygiene practices
  Arms: test mouthrinse
Other: negative control solution — this solution would be used twice per day (2 x 20 ml) following daily home care.
  Arms: control group

SUMMARY:
Chronic periodontitis is a common infectious disease characterized by progressive attachment loss and alveolar bone resorption eventually resulting in tooth loss. The ultimate goal of periodontal therapy is to prevent this endpoint. At least when a strict supportive care program is implemented following active therapy, subsequent tooth loss is limited to a mean of about 0.1 per patient per year. In contrast, three to six times as many teeth may be lost if the disease is left untreated.

The objective of supportive care is to prevent disease recurrence, which is accomplished by strict home care and professional plaque control at regular intervals depending on the patient's needs. Evidently, not all patients are optimally compliant in terms of plaque control. Therefore, chemical aids could be administered to supplement mechanical plaque removal.

Essential oils solutions containing menthol, thymol, methyl salicylate and eucalyptol as active agents may be more appropriate to supplement daily home care. Clinical studies have shown an additional anti-plaque and anti-gingivitis effect over mechanical plaque control without relevant side effects in healthy subjects and gingivitis patients.

Recently, significant reductions of periodontopathogens in the subgingival biofilm have been shown in periodontitis patients following subgingival irrigation using an essential oils solution. In addition, mouthrinsing on a daily basis seemed to substantially alter the subgingival microflora towards a less pathogenic one in gingivitis and periodontitis patients. Even though these are interesting findings, they should be considered exploratory since they relate to a small number of patients observed for only two weeks.

The goal of the present study was to thoroughly document the clinical and microbiological effects of an essential oils solution used on a daily basis for 3 months as an adjunct to mechanical plaque control measures in a large number of chronic periodontitis patients in supportive care.

ELIGIBILITY:
Inclusion Criteria:

* Presence of at least one 4 mm pocket per quadrant
* Patient in maintenance care for at least one year

Exclusion Criteria:

* Presence of 7 mm pockets or more
* Use of antibiotics within 3 months prior to the study
* Patients undergoing orthodontic therapy
* Patients wearing removable partial dentures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-03 (Actual); Primary Completion 2010-05 (Actual); Study Completion 2015-07-31 (Actual)

PRIMARY OUTCOMES:
Clinical and microbiological effects of an essential oils solution. | at 3 months
  Thoroughly document the clinical and microbiological effects of an essential oils solution used on a daily basis for 3 months as an adjunct to mechanical plaque control measures in a large number of chronic periodontitis patients in supportive care.
  These effects are recorded, at baseline (prior to supportive treatment) and after 3 months (again prior to supportive treatment) by the same calibrated clinician

SECONDARY OUTCOMES:
Location of the gingival margin in relation to the cement-enamel junction measured to the nearest mm at 6 sites per tooth using a manual probe | at 3 months
Probing Pocket Depth measured to the nearest mm at 6 sites per tooth using a manual probe. | at 3 months
Bleeding on Probing evaluated 15 seconds following pocket probing | at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Hugo De Bruyn, PhD, Principal Investigator — University Hospital Ghent, Belgium
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: website University Hospital Ghent, Belgium — http://www.uzgent.be